CLINICAL TRIAL: NCT01834235
Title: A Multicenter Phase I/II Randomized Phase II Study of Gemcitabine and Nab-Paclitaxel With or Without NPC-1C in Patients With Metastatic or Locally Advanced Pancreatic Cancer Previously Treated With FOLFIRINOX
Brief Title: QUILT-3.010: A Study of Gemcitabine and Nab-paclitaxel With or Without NPC-1C to Treat Patients With Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: DSMB terminated the trial for futility.
Sponsor: Precision Biologics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PB1201
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer, Adult
Keywords: Pancreatic neoplasms; Pancreatic cancer; Pancreatic cancer, adult; Adenoma of the pancreas; Carcinoma of the pancreas
MeSH Terms: conditions — Pancreatic cancer, adult; Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; ensituximab

STUDY DESIGN:
Intervention Model Description: Initial Phase 1 dose de-escalation design to determine the safe dose of NEO-102 in combination with gemcitabine. Then a Phase 2 randomized design to evaluate the safety and efficacy of gemcitabine and abraxane with or without NEO-102.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Abraxane, gemcitabine (Active Comparator): Nab-paclitaxel will be administered at a dose of 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) followed by 1000 mg/m2 gemcitabine as a 30 minute infusion for 3 consecutive weeks followed by a week of rest.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel
- Abraxane, gemcitabine, NPC-1C (Experimental): Nab-paclitaxel will be administered at a dose of 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) followed by 1000 mg/m2 gemcitabine as a 30 minute infusion for 3 consecutive weeks followed by a week of rest.
  Patients on arm B will receive NPC-1C(NEO-102) infusion at a dose of 1.5mg/kg IV on days 1 and 15 of a 4-week cycle. This will be administered 30minutes after completion of the gemcitabine infusion.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: NPC-1C
- Phase 1: Dose Finding Dose level 1 (Experimental): The initial portion of this protocol was a phase 1 (3+3) dose de-escalation design the initial dose of 1.5 mg/kg/dose:
  Gemcitabine was administered at the dose of 1000 mg/m2 by IV infusions over 30 minutes on days 1, 8, and 15 followed in 30 minutes by NPC-1C(NEO-102) infusion at 1.5 mg/kg IV on days 1 and 15 of a 4-week cycle. Three subjects were enrolled on this dose level and all 3 subjects completed without any dose limiting toxicity. This dose was established for the Phase 2 portion of the study. At this time FDA approved the combination of Gemcitabine and Abraxane in this patient population. Hence the Phase 2 portion added Abraxane to the regimen.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: NPC-1C
- Phase 1: Dose Finding Dose level -1 (Experimental): The initial portion of this protocol was a phase 1 (3+3) dose de-escalation design the initial dose of 1.5 mg/kg/dose:
  Gemcitabine was administered at the dose of 1000 mg/m2 by IV infusions over 30 minutes on days 1, 8, and 15 followed in 30 minutes by NPC-1C(NEO-102) infusion at 1 mg/kg IV on days 1 and 15 of a 4-week cycle. No patients were enrolled on this arm because Dose Level 1 was determined to be safe.
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: NPC-1C

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine IV at a dose of 1000mg/m2 on days 1, 8, and 15 of a 4 week cycle.
  Other Names: gemcitabine (Gemzar)
Drug: nab-paclitaxel — Nab-paclitaxel will be administered at a dose of 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) on Days 1, 7 and 15 for a 28 day cycle
  Other Names: Abraxane
Drug: NPC-1C — NPC-1C(NEO-102) infusion at a dose of 1.5mg/kg IV on days 1 and 15 of a 28 day cycle. This will be administered 30 minutes after completion of the gemcitabine infusion.
  Other Names: Ensituximab
  Arms: Abraxane, gemcitabine, NPC-1C; Phase 1: Dose Finding Dose level -1; Phase 1: Dose Finding Dose level 1

SUMMARY:
This was a Phase 1/2 multi-institution prospective open label study in which subjects with metastatic, locally advanced unresectable or recurrent pancreatic cancer who previously received treatment with chemotherapy with FOLFIRINOX or FOLFIRINOX-like regimen received the investigational agent NEO-102 (NPC-1C).

The Phase 1 portion of this study evaluated the safety of NEO-102 in combination with Gemcitabine in a dose de-escalation design with a starting dose of 1.5 mg/kg/dose. If 2 of 6 patients experience DLT, the dose will be de-escalated to 1 mg/kg/dose to evaluate the safety of NEO-102 in combination with Gemcitabine. .

In the Phase 2 portion patients were randomized into one of two arms:

A: NPC-1C with gemcitabine and nab-paclitaxel or B: gemcitabine and nab-paclitaxel

DETAILED DESCRIPTION:
During Part 1 of the study, the safe and tolerable dose of NEO-102 in combination with Gemcitabine will be determined using a dose de-escalation design. The starting dose of NEO-102 is 1.5 mg/kg/dose (Dose level 1). If 2 of 6 patients experience a DLT at the starting dose, the dose of NEO-102 will be de-escalated to 1 mg/kg/dose, and up to 6 patients will be treated at this Dose Level -1. Upon completion of the phase I study up to 90 patients be randomized to one of two arms:

A: Patients will receive NPC-1C(NEO-102) infusion at the safe dose, and nab-paclitaxel (125 mg/m2 as a 30 minute infusion, maximum infusion time not to exceed 40 minutes) followed by gemcitabine (1000 mg/m2 as a 30 minute infusion) for 3 consecutive weeks (on Day 1, 7 and 15 ) followed by a week of rest (for a 28 day cycle).

OR B: Patients will receive on Day 1, 7 and 15 nab-paclitaxel (125 mg/m2 as a 30 minute infusion, maximum infusion time not to exceed 40 minutes) followed by gemcitabine (1000 mg/m2 as a 30 minute infusion) for 3 consecutive weeks (on Day 1, 7 and 15). NPC-1C(NEO-102) infusion at a dose of 1.5mg/kg IV 30 minutes following the completion of the gemcitabine on days 1 and 15 of the 28 day cycle.

ELIGIBILITY:
Inclusion Criteria

* Subjects with recurrent, locally advanced unresectable or metastatic adenocarcinoma of the pancreas who have progressed after primary therapy with FOLFIRINOX or FOLFIRINOX-like regimen or were intolerant of it.
* IHC greater than or equal to 20 percent of tumor on tissue sections must stain with NPC-1C.
* 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have an anticipated life expectancy of greater than 8 weeks.
* Have recovered from any acute toxicity related to prior therapy.
* If female, is post-menopausal, surgically sterilized or willing to use an effective method of contraception for the duration of the study and for 3 months after the end of treatment. If male, has agreed to use barrier method for contraception for the duration of the study and for 3 months after the end of treatment.
* Must be willing to sign a written informed consent.
* Laboratory tests must meet minimum safety requirements

  1. Hemoglobin greater than or equal to 8.5 g/dL (may be receiving supportive therapy)
  2. ANC greater than or equal to 1,500 K/uL
  3. Platelets greater than or equal to 100 K/uL
  4. Total bilirubin less than or equal to 2 mg/dL
  5. ALT/AST less than or equal to 3 times ULN or less than or equal to 5 times ULN in the setting of liver metastases.
  6. Creatinine less than or equal to 1.5 mg/dL or creatinine clearance greater than 40 mL/min/1.73 m2 for patients with creatinine levels above institutional normal, as calculated by the Cockcroft Gault formula.
* Men and women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria

* Have received a second line chemotherapy after progressing on or not tolerating treatment with FOLFIRINOX as a first line. Prior adjuvant/neoadjuvant gemcitabine or gemcitabine-based radiation will not be counted as first line therapy.
* Have known brain metastases.
* Have had any major surgery within four weeks of enrollment.
* Have greater than grade 2 ascites at time of enrollment.
* Have received Gemcitabine for palliative treatment or progressed while receiving it or is within 3 months of completion in the adjuvant setting.
* Have uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Have serious medical or psychiatric illness that could, in the Investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Must not have other invasive malignancies within the past 3 years (with the exception of non-melanoma skin cancers or non-invasive bladder cancer).
* Is pregnant or breast-feeding, since the effects of NPC-1C on the developing human fetus and nursing infants are unknown and potentially harmful, women of child-bearing potential must agree to use adequate contraception (hormonal or double barrier method of birth control or complete abstinence) prior to study entry, for the duration of study participation, and for three months after the last dose of investigational agent.
* Have had any chemotherapy or systemic corticosteroids within 2 weeks of study entry.
* Have acquired, hereditary or congenital immunodeficiencies including cellular immunodeficiencies, hypogammaglobulinemia and dysgammaglobulinemia.
* Have a prior history of a documented hemolytic event.
* Have a history of hypersensitivity to human or mouse antibody products.
* Have a known history of HIV are excluded due to the possibility that Gemcitabine or NPC-1C(NEO-102) may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events with respect to Gemcitabine or NPC-1C(NEO-102).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-04; Primary Completion 2017-03-13 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Arlen, MD, Study Director — Precision Biologics, Inc
Locations (12):
- United States (12):
  - California Pacific Medical Center, San Francisco, California
  - Smilow Cancer Hospital- Yale, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - National Cancer Institute, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beht Isreal Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Huffman BM, Basu Mallick A, Horick NK, Wang-Gillam A, Hosein PJ, Morse MA, Beg MS, Murphy JE, Mavroukakis S, Zaki A, Schlechter BL, Sanoff H, Manz C, Wolpin BM, Arlen P, Lacy J, Cleary JM. Effect of a MUC5AC Antibody (NPC-1C) Administered With Second-Line Gemcitabine and Nab-Paclitaxel on the Survival of Patients With Advanced Pancreatic Ductal Adenocarcinoma: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jan 3;6(1):e2249720. doi: 10.1001/jamanetworkopen.2022.49720. PMID 36602796

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2 Randomization to Arm A: Patients on arm A will receive Nab-paclitaxel at a dose of 125 mg/m2 as a 30 minute infusion followed by 1000 mg/m2 gemcitabine for 3 consecutive weeks followed by a week of rest (treatment on days 1, 8, and 15, during a 28-day cycle. NPC-1C (NEO-102) will be infused 30 minutes after completion of the gemcitabine infusion at a dose of 1.5mg/kg IV on days 1 and 15 of the 28 day cycle.
- Phase 2 Randomization to Arm B: Nab-paclitaxel will be administered at a dose of 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) followed by 1000 mg/m2 gemcitabine as a 30 minute infusion for 3 consecutive weeks followed by a week of rest (treatment on days 1, 8, and 15, during a 28-day cycle).
- Phase 1-Dose Finding - Dose Level 1: Gemcitabine and NPC-1C at 1.5 mg/kg /dose
- Phase 1 Dose Finding - Dose Level -1: Gemcitabine and NPC-1C at 1 mg/kg/dose
Period: Overall Study
Arm/Group | Phase 2 Randomization to Arm A | Phase 2 Randomization to Arm B | Phase 1-Dose Finding - Dose Level 1 | Phase 1 Dose Finding - Dose Level -1
Started | 38 | 40 | 3 | 0
Completed | 38 | 40 | 3 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: NEO-102 Dose level 1 in combination with Gemcitabine was found to be safe and hence the NEO-102 dose did not need to be de-escalated to Dose level -1.
Groups:
- Phase 1 Dose Finding: Dose Level 1: Patients on arm B will receive NPC-1C(NEO-102) infusion at a dose of 1.5mg/kg IV on days 1 and 15 of a 4-week cycle. This will be administered 30minutes after completion of the gemcitabine 1000 mg/m2 as a 30 minute infusion on days 1, 8, and 15 of a 4 week cycle.
- Phase 1 Dose Finding: Dose Level -1: Patients on arm B will receive NPC-1C(NEO-102) infusion at a dose of 1.0 mg/kg IV on days 1 and 15 of a 4-week cycle. This will be administered 30minutes after completion of the gemcitabine 1000 mg/m2 as a 30 minute infusion on days 1, 8, and 15 of a 4 week cycle.
- Arm A: Abraxane, Gemcitabine, NPC-1C: Nab-paclitaxel will be administered at a dose of 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) followed by 1000 mg/m2 gemcitabine as a 30 minute infusion for 3 consecutive weeks followed by a week of rest.
  Patients on arm B will receive NPC-1C(NEO-102) infusion at a dose of 1.5mg/kg IV on days 1 and 15 of a 4-week cycle. This will be administered 30minutes after completion of the gemcitabine infusion.
  Gemcitabine: Gemcitabine IV at a dose of 1000mg/m2 on days 1, 8, and 15 of a 4 week cycle.
  nab-paclitaxel: Nab-paclitaxel will be administered at a dose of 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) on Days 1, 7 and 15 for a 28 day cycle
  NPC-1C: NPC-1C(NEO-102) infusion at a dose of 1.5mg/kg IV on days 1 and 15 of a 28 day cycle. This will be administered 30 minutes after completion of the gemcitabine infusion.
- Arm B: Abraxane, Gemcitabine: Nab-paclitaxel will be administered at a dose of 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) followed by 1000 mg/m2 gemcitabine as a 30 minute infusion for 3 consecutive weeks followed by a week of rest.
  Gemcitabine: Gemcitabine IV at a dose of 1000mg/m2 on days 1, 8, and 15 of a 4 week cycle.
  nab-paclitaxel: Nab-paclitaxel will be administered at a dose of 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) on Days 1, 7 and 15 for a 28 day cycle
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Finding: Dose Level 1 | Phase 1 Dose Finding: Dose Level -1 | Arm A: Abraxane, Gemcitabine, NPC-1C | Arm B: Abraxane, Gemcitabine | Total
Number analyzed (Participants) | 3 | 0 | 38 | 40 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 26 | 24 | 52
  >=65 years | 1 | 0 | 12 | 16 | 29
Age, Continuous [Median (Full Range); unit: years] | 53 [51 to 80] |  | 62 [36 to 78] | 62.5 [37 to 78] | 62 [36 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 19 | 29 | 51
  Male | 0 |  | 19 | 11 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 3 | 4 | 8
  Not Hispanic or Latino | 2 |  | 33 | 34 | 69
  Unknown or Not Reported | 0 |  | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0 | 0
  Asian | 0 |  | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0 | 0
  Black or African American | 2 |  | 4 | 5 | 11
  White | 1 |  | 32 | 34 | 67
  More than one race | 0 |  | 0 | 0 | 0
  Unknown or Not Reported | 0 |  | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 38 | 40 | 81
NPC-1C IHC staining [Number; unit: participants positive] | 3 |  | 38 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: To determine the safety and tolerability of NPC-1C monoclonal antibody therapy in combination with Gemcitabine in subjects with metastatic, locally advanced unresectable or recurrent pancreatic cancer who failed or did not tolerate first line chemotherapy of FOLFIRINOX and whose tumors bind NPC-1C.
Time Frame: 28 days
Population: Dose level -1 did not enroll any patients because dose level 1 was found to be safe when NEO-102 was given in combination with Gemcitabine. Hence there was no need to dose de-escalate.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1-Dose Finding Dose Level 1: Gemcitabine will be administered at the dose of 1000 mg/m2 by IV infusions over 30 minutes on days 1, 8, and 15 followed in 30 minutes by NPC-1C(NEO-102) 1.5 mg/kg infusion on days 1 and 15 of a 4-week cycle.
- Phase 1 Dose Finding: Dose Level -1: Gemcitabine will be administered at the dose of 1000 mg/m2 by IV infusions over 30 minutes on days 1, 8, and 15 followed in 30 minutes by NPC-1C(NEO-102) 1.5 mg/kg infusion on days 1 and 15 of a 4-week cycle. No patients were enrolled to this de-escalated dose because Dose Level 1 was found to be safe when given in combination with Gemcitabine.
- Arm A: Abraxane, Gemcitabine, NPC-1C: Patients on arm A will receive Nab-paclitaxel at a dose of 125 mg/m2 as a 30 minute infusion followed by 1000 mg/m2 gemcitabine for 3 consecutive weeks followed by a week of rest (treatment on days 1, 8, and 15, during a 28-day cycle. NPC-1C (NEO-102) will be infused 30 minutes after completion of the gemcitabine infusion at a dose of 1.5mg/kg IV on days 1 and 15 of the 28 day cycle.
- Arm B: Abraxane, Gemcitabine: Nab-paclitaxel will be administered at a dose of 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) followed by 1000 mg/m2 gemcitabine as a 30 minute infusion for 3 consecutive weeks followed by a week of rest (treatment on days 1, 8, and 15, during a 28-day cycle).
Arm/Group | Phase 1-Dose Finding Dose Level 1 | Phase 1 Dose Finding: Dose Level -1 | Arm A: Abraxane, Gemcitabine, NPC-1C | Arm B: Abraxane, Gemcitabine
Number analyzed (Participants) | 3 | 0 | 38 | 40
Participants | 0 |  | 3 | 7

2. Primary Outcome: Overall Survival
Description: To determine whether (only in participants in the Phase 2 portion (Arm A and Arm B) NPC-1C (NEO-102) in combination with Gemcitabine and nab-Paclitaxel will increase the overall survival (OS) compared to Gemcitabine and nab-Paclitaxel alone in patients with metastatic, locally advanced unresectable or recurrent pancreatic cancer previously treated with FOLFIRINOX and whose tumors bind NPC-1C by at least 20% on IHC.
Time Frame: From 1st dose of study therapy until death in participants in Phase 2.
Population: 78 participants who received study therapy in the Phase 2 portion of the study. Patients in the Phase 1 portion of the study were not included in the Analysis of outcome measure #2 because they only received NPC-1C and Gemcitabine.
Measure: Median (95% Confidence Interval); unit: Number of months survival
Arm/Group | Arm A: Abraxane, Gemcitabine, NPC-1C | Arm B: Abraxane, Gemcitabine
Number analyzed (Participants) | 38 | 40
Number of months survival | 6.6 [4.7 to 8.4] | 5 [3.3 to 6.5]

3. Secondary Outcome: Progression Free Survival
Description: To determine the progression free survival (PFS) and response rate (RR) of patients with metastatic or locally advanced unresectable or recurrent pancreatic cancer who progressed following or did not tolerate chemotherapy of FOLFIRINOX or FOLFIRINOX-like regimen when receiving the combination of NPC-1C(NEO-102) monoclonal antibody, Gemcitabine and nab-Paclitaxel (Arm A).
Time Frame: Time from the 1st dose of study drug until progression in patients in Arm A
Population: 78 participants who received study therapy in the Phase 2 portion of the study. Patients in the Phase 1 portion of the study were not included in the Analysis of outcome measure #3 because they only received NPC-1C and Gemcitabine.
Measure: Median (95% Confidence Interval); unit: Median number of months without PD
Groups:
- Arm A: Patients on arm A will receive Nab-paclitaxel at a dose of 125 mg/m2 as a 30 minute infusion followed by 1000 mg/m2 gemcitabine for 3 consecutive weeks followed by a week of rest (treatment on days 1, 8, and 15, during a 28-day cycle. NPC-1C (NEO-102) will be infused 30 minutes after completion of the gemcitabine infusion at a dose of 1.5mg/kg IV on days 1 and 15 of the 28 day cycle.
- Arm B: Nab-paclitaxel will be administered at a dose of 125 mg/m2 as a 30 minute infusion (maximum infusion time not to exceed 40 minutes) followed by 1000 mg/m2 gemcitabine as a 30 minute infusion for 3 consecutive weeks followed by a week of rest (treatment on days 1, 8, and 15, during a 28-day cycle).
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 38 | 40
Median number of months without PD | 3.5 [2.0 to 5.6] | 2.7 [1.9 to 4.1]

ADVERSE EVENTS:
Time Frame: Through study completion an average of 8 months
Description: A event is considered serious if it results in any of the following:
  * Death,
  * A life-threatening AE
  * Inpatient hospitalization or prolongation
  * Persistent or significant incapacity
  * A congenital anomaly/birth defect.
  * Important medical events that may not result in death, be life-threatening, or require hospitalization
Groups:
- Phase 1- Dose Finding -Dose Level 1: Gemcitabine and NPC-1c at 1.5 mg/kg/dose
- Phase 1- Dose Finding -Dose Level -1: Gemcitabine and NPC-1c at 1.0 mg/kg/dose
Arm/Group | Arm A | Arm B | Phase 1- Dose Finding -Dose Level 1 | Phase 1- Dose Finding -Dose Level -1
All-Cause Mortality (participants affected / at risk) | 38/38 | 40/40 | 3/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 18/38 | 12/40 | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 32/38 | 33/40 | 0/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=38) | Arm B (N=40) | Phase 1- Dose Finding -Dose Level 1 (N=3) | Phase 1- Dose Finding -Dose Level -1 (N=0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA | NA
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 2 (2) | NA | NA
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 4 (4) | NA | NA
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA | NA
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | NA | NA
Neutrophil Count Decreased (Investigations) | 2 (2) | 0 (0) | NA | NA
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA | NA
Aspartate Aminotransferase increased (Investigations) | 1 (1) | 0 (0) | NA | NA
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Infection lung (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Infection Urinary Tract (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | NA | NA
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA | NA
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=38) | Arm B (N=40) | Phase 1- Dose Finding -Dose Level 1 (N=3) | Phase 1- Dose Finding -Dose Level -1 (N=0)
Absolute Lymphocyte count decreased (Investigations) | 3 (8) | 3 (4) | NA | NA
Alkaline Phosphatase increased (Investigations) | 4 (4) | 0 (0) | NA | NA
Anemia (Blood and lymphatic system disorders) | 15 (22) | 4 (7) | NA | NA
Fatigue (General disorders) | 5 (5) | 1 (2) | NA | NA
Neutropenia (Investigations) | 13 (15) | 12 (16) | NA | NA
Platelet count decreased (Investigations) | 12 (13) | 8 (13) | NA | NA
White blood cell count decreased (Investigations) | 9 (9) | 5 (5) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT01834235/Prot_SAP_000.pdf